CLINICAL TRIAL: NCT04300829
Title: Randomised Multicentric Phase III Study Evaluating the Efficacy of Cicaderma vs Standard Management of Each Site in Preventing Radiodermatitis After Adjuvant Post-operative Breast Irradiation in Patients With Non-metastatic Breast Cancer
Brief Title: Cicaderma Efficacy vs Standard Care of Sites in Preventing Radiodermatitis in Non-metastatic Breast Cancer Patients
Acronym: CICA-RT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET19-084 - CICA-RT
Record Dates: First submitted 2020-02-28; First posted 2020-03-09 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Breast Adenocarcinoma; Radiation Dermatitis; Radiation Toxicity
Keywords: Non-metastatic breast cancer; Post operative adjuvant radiotherapy; Radiotherapy cutaneous toxicity
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, multicentric Phase III study evaluating the Cicaderma ointment efficacy versus standard practice of each site in the prevention of radiodermatitis in patients presenting a non metastatic breast cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple hygiene rules of the site + Cicaderma ointment (Experimental): Hygiene rules (use of a neutral soap, no bath, use of non-alcoholic products, delicate drying of the skin, wearing of cotton clothing) and Cicaderma ointment application)
  Interventions: Drug: cicaderma + simple hygiene rules
- Preventive standard cares (Active Comparator): Preventive standard cares of the site including hygiene rules (use of a neutral soap, no bath, use of non-alcoholic products, delicate drying of the skin, wearing of cotton clothing) and a maximum of one topical treatment
  Interventions: Other: Simple hygiene rules and a maximum of one topical treatment

INTERVENTIONS:
Drug: cicaderma + simple hygiene rules — Cicaderma ointment (2 applications / day: after the radiotherapy session) and in the evening) + simple hygiene rules
  Other Names: Cicaderma ointment and simple hygiene rules
  Arms: Simple hygiene rules of the site + Cicaderma ointment
Other: Simple hygiene rules and a maximum of one topical treatment — Simple hygiene rules according to the site recommandations including eventually a maximum of one topical treatment
  Arms: Preventive standard cares

SUMMARY:
Phase III, prospective, interventional, multicentric, comparative, randomized, open study with 2 parallel arms, evaluating the efficacy of Cicaderma ointment vs standard management of each site in preventing the onset of grade > 2 radiodermatitis according to the National Cancer Institute - Common Terminology Criteria for Adverse Events-Version (NCI-CTCAE-V5)

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. It accounts for more than 1/3 of new cancer cases and is the 1st cause of death for women.

Management usually includes tumorectomy or mastectomy precede or not by a chemotherapy, then adjuvant irradiation that can be supplemented with adjuvant chemotherapy and / or hormone therapy.

Radiotherapy uses ionizing radiation (photons, electrons ...) to destroy cancer cells and consists in precisely directing these radiations on the area to be treated while preserving as much as possible healthy tissues and surrounding organs.

Radiation-induced dermatitis is a skin lesion that occurs after exposure to ionizing radiation and is commonly seen in patients. Acute radiodermatitis occurs in the days or weeks following the start of irradiation with different degrees of severity (dry or exsudative radiodermatitis, acute radionecrosis) They are responsible for an alteration of patients' quality of life (pain, sensitivity to UV radiation, discomfort sensations ...), which may lead to a temporary or even permanent therapeutic interruption and reduce the probability of tumor control.

The management of these dermatitis is very heterogeneous, no study having demonstrated the superiority of a preventive or curative treatment. Trolamine (Biafine®) is to date the only topic with a Marketing Authorization (MA) for the treatment of radiation-induced secondary erythema.

A study conducted on 254 patients at the Léon Bérard Center from 1999 to 2001 demonstrated that the preventive use of a calendula-based topical was associated with a statistically significant reduction of grade 2 radiodermitis compared to trolamine in patients presenting an early breast cancer treated with post-operative irradiation. However, this calendula ointment, which does not have the MA in the indicated indication, was in practice more difficult to apply than trolamine.

Currently, skin hygiene measures to be applied are systematically explained to patients before carrying out post-operative radiotherapy (cotton clothing, neutral soap, etc.). Some centers such as Center Léon Bérard recommend the systematic use of a topic after each session, while others recommend hygiene measures or implement other options (essential oils ...). However, the effectiveness of these current practices on the prevention of radiodermatitis has not yet been demonstrated.

It is a phase III, prospective, interventional, multicentric, comparative, randomized, open study with 2 parallel arms Patients will be randomized (1 :1) in Arm A (hygiene measures + preventive treatment with Cicaderma ointment) or Arm B (preventive treatment according to the site recommendations (at least the hygiene measures) with a stratification (site, body mass index ≤25 vs >25 and RT hypofractionning).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient requiring a post-operative radiotherapy (post mastectomy or tumorectomy) for a mammary adenocarcinoma or an unilateral in situ breast cancer histologically documented, early stage of disease (non metastatic)
* Patient with no residual tumor (R0 or R1)
* Patient informed and having given her signed consent
* Patient affiliated to a social security regimen

Exclusion Criteria:

* Unsolved cutaneous toxicities of any previous treatment
* Hormonotherapy started prior to radiotherapy
* Concomitant use of other topical treatments than the study treatments on the irradiated area
* Patient treated by concomitant chemotherapy and/or targeted therapy
* Known hypersensibility to at least one component of the topicals used or Cicadema ointment
* Patient for whom follow-up does not seem possible even in the short term
* Pregnant or breastfeeding woman
* Participation in another clinical trial that may interfere with the evaluation of the primary endpoint
* Patient Under tutorship or curatorship or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-09-09 (Estimated); Study Completion 2022-10-09 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Cicaderma ointment efficacy versus the standard management of each site in preventing the onset of grade >= 2 radiodermatitis (NCI-CTCAE-V5) | Up to 30+/-4 days after the end of radiotherapy interruption
  Number of patients presenting >= 2 radiodermatitis according to the National Cancer Institute - Common Terminology Criteria for Adverse Events-Version (NCI-CTCAE-V5)

SECONDARY OUTCOMES:
Patients' satisfaction | 30+/-4 days after the end of radiotherapy interruption
  Patients' satisfaction evaluated using the "Patient's evaluation of the preventive management of radiodermatits" - Likert scale in 5 points (from very unsatisfied to very satisfied)
Patients' quality of life: DLQI questionnaire | Up to 30+/-4 days after the end of radiotherapy interruption
  Patients' quality of life evaluated using the Dermatology Life Quality Index (DLQI) questionnaire (validated questionnaire composed of 10 items leading to a global score)
Patients' pain in the irradiated area: numeric scale | Up to 30+/-4 days after the end of radiotherapy interruption
  Patients' pain evaluated using a numeric scale from 0 (no pain) to 10 (unbearable pain)
Rate of temporary or permanent RT interruption related to the onset of grade 3 radiodermatitis | Through radiotherapy completion, an average of 5 weeks
  Temporary or permanent radiotherapy interruption related to the onset of grade 3 radiodermatitis observed during patients' treatment period
Rate of prurit onset whatever the grade | Up to 30+/-4 days after the end of radiotherapy interruption
  Prurit onset whatever the grade observed
Doses of radiation therapy received | Through radiotherapy completion, an average of 5 weeks
  Doses of radiation therapy received during each radiotherapy session
Delay of onset of the first cutaneous event (radiodermatitis or prurit) grade ≥2 | Up to 30+/-4 days after the end of radiotherapy
  Onset of the first grade >= 2 cutaneous event (radiodermatitis or prurit)
Compliance with the Cicaderma ointment application (experimental arm) | Up to 30+/-4 days after the end of radiotherapy
  Compliance evaluated according to the ointment tubes brought back by the patients (not used or partially used) and patient's diary
Determination of the factors measured prior to treatment initiation which are associated to the onset of grade ≥2 radiodermatitis (cup size) | At inclusion
  Cup size
Determination of the factors measured prior to treatment initiation which are associated to the onset of grade ≥2 radiodermatitis (phototype) | At inclusion
  Phototype

CONTACTS AND LOCATIONS:
Overall Officials: Séverine RACADOT, MD, Principal Investigator — Centre Leon Berard; Youlia KIROVA, MD PhD, Principal Investigator — Institut Curie
Locations (3):
- France (3):
  - Institut Sainte-Catherine, Avignon
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

REFERENCES:
- [Derived] Racadot S, Arnaud A, Schiffler C, Metzger S, Perol D, Kirova Y. Cicaderma(R) in radiation-related dermatitis of breast cancer: Results from the multicentric randomised phase III CICA-RT. Clin Transl Radiat Oncol. 2023 Jun 1;41:100647. doi: 10.1016/j.ctro.2023.100647. eCollection 2023 Jul. PMID 37441546